CLINICAL TRIAL: NCT03093259
Title: Phase IIa Study to Evaluate the Safety and Efficacy of ABX464 Versus Placebo in Subjects With Moderate to Severe Active Ulcerative Colitis Who Have Failed or Are Intolerant to Immunomodulators, Anti-TNFα, Vedolizumab and/or Corticosteroids
Brief Title: ABX464 in Subjects With Moderate to Severe Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABX464-101
Record Dates: First submitted 2017-03-17; First posted 2017-03-28 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis
Keywords: ABX464; Ulcerative Colitis; Refractory
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ABX464

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind Treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABX464 Treatment Arm (Experimental): Subjects will receive 50 mg of ABX464 orally once daily for 56 days.
  Interventions: Drug: ABX464
- ABX464 matching placebo Treatment Arm (Placebo Comparator): Subjects will receive 50 mg of ABX464 matching Placebo orally once daily for 56 days.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ABX464 — ABX464 is a new Anti-inflammatory drug
  Arms: ABX464 Treatment Arm
Drug: Placebo oral capsule — Placebo matching with ABX464
  Arms: ABX464 matching placebo Treatment Arm

SUMMARY:
This Phase IIa study is an 8-week, double-blind, placebo-controlled, randomized study aiming at evaluating the safety and the efficacy of ABX464 given once a day (o.d) at 50 mg in subjects with moderate to severe Active Ulcerative Colitis who have failed or are intolerant to immunomodulators, Anti-TNFα, vedolizumab and/or corticosteroids followed by a one-month follow-up period.

DETAILED DESCRIPTION:
This Phase IIa study is an 8-week, double-blind, placebo-controlled, randomized study aiming at evaluating the safety and the efficacy of ABX464 given once a day (o.d) at 50 mg in subjects with moderate to severe Active Ulcerative Colitis who have failed or are intolerant to immunomodulators, Anti-TNFα, vedolizumab and/or corticosteroids followed by a one-month follow-up period.

Eligible subjects will be randomized according to a 2/1 ratio in two different groups of treatment. Randomized subjects who will receive 50 mg ABX464 orally once daily for 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe active UC confirmed by endoscopy and histology at least 12 weeks prior to screening visit. Moderate to severe active UC defined by Mayo Clinic Score (MCS) of 6 to 12 inclusive (on a scale of 0-12). Moderate to severe active UC should be confirmed at screening visit with a centrally read MCS endoscopy score of at least 2 (on a scale of 0-3);
* Subjects receiving oral corticosteroids must have been on a stable dose of prednisone or prednisone equivalent ≤20 mg/day) or on beclomethasone diproprionate (≤5mg/day) or on budesonide MMX (≤9mg/day), for ≥2 weeks before first dosing (i.e. baseline);
* Topical corticosteroids and topical 5-aminosalicylic acid preparations must have been withdrawn ≥2 weeks before first dosing (i.e. baseline);
* Subjects who are on oral 5-aminosalicylic acid must have been on a stable dose ≥4 weeks before first dosing (i.e. baseline);
* Subjects who are receiving immunosuppressants in the form of azathioprine, 6-mercaptopurine, or methotrexate needed to be on a stable dose for 4 weeks before first dosing (i.e. baseline). Subjects taking methotrexate also are advised to take folic acid 1 mg/day (or equivalent) supplementation if there is no contraindication;
* Subjects on probiotics (e.g., Culturelle® [Lactobacillus GG, i-Health, Inc.], Saccharomyces boulardii) must be on stable doses for 2 weeks before first dosing (i.e. baseline);
* Subjects on antidiarrheals (e.g., loperamide, diphenoxylate with atropine) must be on stable doses for 2 weeks before first dosing (i.e. baseline);
* Subjects who have previously received anti-tumor necrosis factor (TNF) therapy or vedolizumab must have discontinued therapy ≥8 weeks before first dosing (i.e. baseline);
* Subjects previously treated with cyclosporine or tacrolimus must have discontinued therapy ≥4 weeks before first dosing (i.e. baseline);
* Subjects previously treated with tube feeding, defined formula diets, or parenteral alimentation/nutrition must have discontinued treatment 3 weeks before first dosing (i.e. baseline).

Exclusion Criteria:

* Subject with Crohn's Disease (CD), indeterminate colitis (IC) or presence or history of fistula with CD;
* History of toxic megacolon, abdominal abscess, symptomatic colonic stricture or stoma; history or is at imminent risk of colectomy;
* History or current evidence of colonic dysplasia or adenomatous colonic polyps. Subject with severe gastrointestinal complications; e.g., short bowel syndromes, obstructing strictures, recent or planned bowel surgery, Ileostomy and/or colostomy, recent bowel perforation;
* Subject with significant and known active infections at screening such as Infected abscess, positive for Clostridium difficile (stool antigen and toxin), CMV, TB and recent infectious hospitalization;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Univ.-Klinik für Innere Medizin I, Innsbruck, Austria
- University Hospitals Leuven - campus Gasthuisberg, Leuven, Belgium
- Czechia (2):
  - Klinické centrum ISCARE, Prague
  - Orlicko-ustecka nemocnice, Ústí nad Orlicí
- France (4):
  - CHRU de Lille, Lille
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHU Saint Etienne - CHU Hopital Nord, Saint-Priest-en-Jarez
- Germany (2):
  - Medizinische Klinik für Gastroenterologie, Infektiologie und Rheumatologie, Berlin
  - Akademisches Lehrkrankenhaus Christian-Albrechts-Universität zu Kiel, Hamburg
- Hungary (3):
  - DRC Gyógyszervizsgáló Központ Kft, Balatonfüred
  - Belgyógyászati Klinika, Budapest
  - Vasútegészségügyi Nonprofit Közhasznú Kft.,, Debrecen
- Poland (5):
  - Centrum Badań, Lodz
  - KO-Med, Lublin
  - Medpolonia Poznań, Poznan
  - NZOZ ViVamed, Warsaw
  - Centrum Badań Klinicznych Lekarze Sp.p, Wroclaw
- Hospital RAMÓN Y CAJAL, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABX464 Treatment Arm | ABX464 Matching Placebo Treatment Arm
Started | 23 | 9
Completed | 21 | 9
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of ABX464.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABX464 Treatment Arm | ABX464 Matching Placebo Treatment Arm | Total
Number analyzed (Participants) | 23 | 9 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 9 | 28
  >=65 years | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 1 | 12
  Male | 12 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 23 | 9 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events
Description: Number of treatment-emergent adverse events in the ABX464 treated subjects compared to placebo
Time Frame: Week 8
Population: All subjects who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 Treatment Arm | ABX464 Matching Placebo Treatment Arm
Number analyzed (Participants) | 23 | 9
Participants | 18 | 5
Statistical Analysis 1: Comparison: ABX464 Treatment Arm vs ABX464 Matching Placebo Treatment Arm; Test type: Other — One-sided 10% significance level; p = 0.2096, Chi-squared

2. Secondary Outcome: Clinical Remission
Description: Percentage of subjects receiving ABX464 with clinical remission according to the Total Mayo Score at Week 8 compared to placebo (primary efficacy endpoint)
Time Frame: Week 8
Population: Subjects in the FAS without any major protocol deviations and who completed the study (Day 56)
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 Matching Placebo Treatment Arm | ABX464 Treatment Arm
Number analyzed (Participants) | 20 | 9
Participants | 7 | 1
Statistical Analysis 1: Comparison: ABX464 Matching Placebo Treatment Arm vs ABX464 Treatment Arm; Test type: Other; p = 0.1588, Chi-squared

3. Secondary Outcome: Fecal Calprotectin
Description: Percentage of patients with fecal calprotectin levels > 50µg/g at Week 8 compared to placebo
Time Frame: Week 8
Population: Subjects in the FAS without any major protocol deviations and who completed the study (Day 56)
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 Treatment Arm | ABX464 Matching Placebo Treatment Arm
Number analyzed (Participants) | 20 | 9
Participants | 15 | 8
Statistical Analysis 1: Comparison: ABX464 Treatment Arm vs ABX464 Matching Placebo Treatment Arm; Test type: Other; p = 0.4830, ANCOVA

4. Secondary Outcome: Total Mayo Score
Description: Change from baseline in Total Mayo Score in subjects receiving ABX464 compared to placebo. The scale ranges from 0 to 12; 12 being the worst score) - 4-component Scale: Rectal bleeding, Stool frequency, Mucosal appearance and Physician Global Assessment
Time Frame: Week 8
Population: Subjects in the FAS without any major protocol deviations and who completed the study (Day 56)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABX464 Treatment Arm | ABX464 Matching Placebo Treatment Arm
Number analyzed (Participants) | 20 | 9
score on a scale | -4.6 (2.8) | -2.1 (2.5)
Statistical Analysis 1: Comparison: ABX464 Treatment Arm vs ABX464 Matching Placebo Treatment Arm; Test type: Other; p = 0.0742, ANCOVA

5. Secondary Outcome: Change in Partial Mayo Score
Description: Change from baseline in Partial Mayo Score in subjects receiving ABX464 compared to placebo. The scale ranges from 0 to 9, with 9 indicating the worst score. It is a three-component scale assessing rectal bleeding, stool frequency, and the physician's global assessment.
Time Frame: Week 8
Population: Subjects in the FAS without any major protocol deviations and who completed the study (Day 56)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABX464 Treatment Arm | ABX464 Matching Placebo Treatment Arm
Number analyzed (Participants) | 20 | 9
units on a scale | -3.9 (2.2) | -1.8 (2.0)
Statistical Analysis 1: Comparison: ABX464 Treatment Arm vs ABX464 Matching Placebo Treatment Arm; Test type: Other; p = 0.0462, ANCOVA

ADVERSE EVENTS:
Time Frame: From baseline up to 4 weeks post last dose of study drug (up to 63 Days)
Description: During the study, in case of a safety evaluation, the investigator or site staff will be responsible for reporting AEs and SAEs, as detailed in this section of the protocol. Participants may report AEs occurring at any other time during the study.
Groups:
- ABX464: Participants received 1 oral capsule containing ABX464 daily for 56 days
- Placebo: Participants received 1 oral capsule containing placebo daily for 56 days
Arm/Group | ABX464 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/9
Other Adverse Events (participants affected / at risk) | 18/23 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 (N=23) | Placebo (N=9)
Nephrolithiasis left side (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABX464 (N=23) | Placebo (N=9)
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Influenza like illness (General disorders) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
AST/ALT ratio (Investigations) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT03093259/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT03093259/SAP_001.pdf